CLINICAL TRIAL: NCT02293720
Title: An Open-Label Extension to Protocol 09-1, Multi-Center, Efficacy and Safety Study of the EndoBarrier® Gastrointestinal Liner System for Glycemic Improvement in Inadequately Controlled Obese Type 2 Diabetic Subjects
Brief Title: An Open-Label Extension to Protocol 09-1, Efficacy and Safety Study of the EndoBarrier® Gastrointestinal Liner System
Acronym: OLE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This was the cross over study for 09-1 which was terminated early
Sponsor: Morphic Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-1E
Record Dates: First submitted 2014-11-11; First posted 2014-11-18 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2014-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EndoBarrier Device (Experimental): Subjects who participated in the control arm of study #09-1 who are not treatment failures and have completed 12 months of the study. These subjects will have the EndoBarrier device implanted for 12 months.
  Interventions: Device: EndoBarrier

INTERVENTIONS:
Device: EndoBarrier — The EndoBarrier is indicated as an adjunct to diet and exercise to achieve weight loss and improve glycemic control in obese adults with type 2 diabetes whose anti-diabetes medications have not achieved adequate glycemic control.

SUMMARY:
A multi-center, single-arm, open-label study to evaluate the safety and effectiveness of the EndoBarrier Gastrointestinal Liner System liner on glycemic control in control subjects from study #09-1 who are not treatment failures and have completed 12 months of the study.

DETAILED DESCRIPTION:
This is an open-label extension study for subjects who participated in the control arm of study #09-1 (A Randomized, Multi-Center, Pivotal Efficacy and Safety Study Comparing the EndoBarrier Gastrointestinal Liner System vs. Sham for Glycemic Improvement in Inadequately Controlled Obese Type 2 Diabetic Subjects on Oral Anti-Diabetes Agents) who are not treatment failures and completed 12 months of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Control subjects from study # 09-1 who are not treatment failures and have completed 12 months of the study
2. Age ≥21 years and ≤ 65 years
3. Have signed an informed consent form within 30 days of week 52 visit in study #09-1.
4. HbA1c ≥ 7.5% and ≤ 10%
5. Stable (s) doses (up to 2) of anti -diabetes medication(s) for a minimum of 3 months prior to enrollment with at least one at minimum required dose as outlined below:

   1. MET (≥1500 mg/day) OR
   2. SU (based on doses specified below) Generic Name (brand name) minimum required dose

      Glimepiride (Amaryl) 4 (mg/day) Glipizide (Glucotrol) 20 (mg/day) Glipizide (Glucotrol XL) 10 (mg/day) Glyburide (Micronas, Diabeta) 10 (mg/day) Micronized Glyburide (Glynase) 6 (mg/day) Chlorpropamide (Diabinese) 350 (mg/day) Tolazamide (Tolinase 500 (mg/day) Tolbutamide (Orinase) 1500 (mg/day) OR
   3. DPP-4i (based on doses specified below) Generic Name (brand name) minimum required dose Sitagliptin (Januvia®) 50 (mg/day) Saxagliptin (Onglyza®) 2.5 (mg/day) Linagliptin (Tradjenta ®) 5 (mg/day) Alogliptin (Nesina®) 12.5 (mg/day)
   4. TZD (based on doses specified below) Generic Name (brand name) minimum required dose Rosiglitazone (Avandia®) 4 (mg/day) Pioglitazone (Actos®) 30 (mg/day)
6. BMI ≥ 30 and ≤ 55
7. Willing to comply with study requirements
8. Documented negative pregnancy test in women of childbearing potential
9. Women of childbearing potential not intending to become pregnant for the duration of their trial participation

Exclusion Criteria

1. Any change from the subject's previous health status from assessment for eligibility in pivotal trial phase (such as a new condition or major illness) that places the subject at undue risk by participating in the study
2. C-peptide < 1.0 ng/mL
3. Triglyceride level > 400 mg/dL
4. Vitamin D deficiency (<20ng/ml)
5. Male subjects with serum Cr >1.5 mg/dl or female subjects with Cr >1.4 mg/dl
6. Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 100,000/microliter, or known coagulopathy
7. Symptomatic kidney stones or gallstones within 6 months prior to baseline (within 30 days of week 52 visit from #09-1 study)
8. Acute pancreatitis at the time of baseline (within 30 days of week 52 visit from #09-1 study)
9. Diagnosis of osteoporosis or currently taking bisphosphonates or teriparatide
10. Currently taking Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) (e.g. aspirin, ibuprofen, etc.) within 10 days of the procedure and/or there is a need or expected need to use during the trial 12 months post index procedure
11. Currently taking prescription antithrombotic therapy (e.g. anticoagulant or antiplatelet agent) within 10 days prior to the procedure and/or there is a need or expected need to use during the trial 12 months post index procedure
12. Currently taking the following medications (at the time of enrollment) and/or there is a need or expected need to use these medications during the trial 12 months post index procedure:

    Restricted Medications/Supplements Systemic corticosteroids Drugs known to affect GI motility (e.g. Reglan) Prescription or over-the-counter weight loss medication(s) Medications known to cause significant weight gain (refer to study reference manual (SRM) or weight loss (e.g. chemotherapeutics)
13. Currently taking ≥ two of the following medications for type 2 diabetes; MET, SU, DDP-4i and TZD at baseline (within 30 days of week 52 visit from #09-1 study)
14. Currently taking medications for type 2 diabetes other than MET, SU, DPP-4i, and TZD (e.g. GLP1 or insulin) at baseline (within 30 days of week 52 visit from #09-1 study)
15. Chronic use of narcotics, opiates, or benzodiazepines and other addictive tranquilizers
16. Allergy or hypersensitivity to ceftriaxone, cephalosporins, penicillin, and all equivalent antibiotics
17. Active H. pylori (Note: Subjects may be eligible after undergoing 2 weeks of antibiotic treatment without re-screening)
18. Residing in a location without ready access to study site medical resources
19. Documented weight loss of > 10 pounds anytime during the 3 months prior to enrollment

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Mean change in HbA1c value from baseline to 12 months | 52 weeks
  Changes in HbA1c from baseline to 12 month
Measure the incidence of device related serious adverse events requiring an early removal | 52 weeks
  Demonstrated to be less than or equal to 15%

IPD SHARING:
Plan to Share IPD: No